CLINICAL TRIAL: NCT06011382
Title: Maxillary Molar Distalization Supported by Mini-implants With the Advanced Molar Distalization Appliance (Amda®): A Randomized Controlled Trial
Brief Title: Maxillary Molar Distalization Supported by Mini-implants With the Advanced Molar Distalization Appliance (Amda®)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grigore T. Popa University of Medicine and Pharmacy (Other)
Collaborators: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Nikolaos Karvelas, Principal Investigator, Grigore T. Popa University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NKarvelas
Record Dates: First submitted 2023-06-13; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Angle Class II
Keywords: amda®; maxillary molar distalization; randomized controlled trial; orthodontics
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Intervention Model Description: Two arm parallel randomized controlled trial with 1:1 allocation ratio
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- patients treated with amda® (Active Comparator): two different treatment groups will be evaluated, from initiation of treatment until completion of maxillary molar distalization.
  Interventions: Device: Advanced Molar Distalization Appliance (amda®)
- patients treated with buccal mini-implants (Active Comparator): from initiation of treatment until completion of maxillary molar distalization.
  Interventions: Device: Buccal mini-implants

INTERVENTIONS:
Device: Advanced Molar Distalization Appliance (amda®) — AMDA is a prefabricated device anchored to the palate by miniscrews and it is a noncompliance appliance for maxillary molar distalization
  Arms: patients treated with amda®
Device: Buccal mini-implants — Buccal mini-implants for maxillary molar distalization
  Arms: patients treated with buccal mini-implants

SUMMARY:
The aim of this randomized controlled clinical trial is to evaluate the dentoalveolar and skeletal treatment effects of the AMDA when used for distalization of the maxillary first molars in patients with Class II malocclusion in the permanent dentition.

DETAILED DESCRIPTION:
The primary aim is to evaluate two different treatment groups from initiation of treatment up until completion of maxillary molar distalization of:

* Group I: patients treated with amda®
* Group II: patients treated with buccal mini-implants

More specifically to evaluate the efficiency of the AMDA using lateral cephalograms and digital 3D model casts of the patients under investigation at the following time points:

* point T0: baseline data - before initiation of the treatment
* point T1: immediately after distalization (8-12 months)

ELIGIBILITY:
Inclusion Criteria:

* All patients to have permanent dentition
* with or without the 2nd molar erupted
* bilateral Class II molar relationships (a quarter to 1 molar cusp).

Exclusion Criteria:

* Past orthodontic treatment
* crossbites,
* severe carious lesions,
* poor oral hygiene,
* mobility of the maxillary first molars,
* anterior open bites,
* vertical growth pattern,
* tongue habits.

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2024-06-20 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Anteroposterior position changes of upper first molars. | 8-12 months
  Anteroposterior position movement in mm of the upper first molars
Measurements on the lateral cephalograms and digital 3D model casts. | 8-12 months
  Angular measurements of the lateral cephalograms and digital models
Measurements on the lateral cephalograms and digital 3D model casts. | 8-12 months
  Linear measurements of the lateral cephalograms and digital models

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Karvelas, PhD student, Principal Investigator — Grigore T Popa University, Department of Orthodontics
Locations (1):
- University of Medicine and Pharmacy "Grigore T. Popa", Iași, Romania

IPD SHARING:
Plan to Share IPD: No
The data will be availaible upon request